CLINICAL TRIAL: NCT00945425
Title: A Phase I, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD7325 When Given in Multiple Ascending Oral Doses in Healthy Male Japanese Subjects
Brief Title: AZD7325 Japan Multiple Ascending Dose (MAD) Study
Acronym: JMAD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decided to stop development of this compound globally
Sponsor: AstraZeneca (Industry)
Responsible Party: Raj Tummala, MD-Medical Science Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D1140C00015
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: Phase I; Volunteer
MeSH Terms: interventions — 4-amino-8-(2-fluoro-6-methoxy-phenyl)-N-propylcinnoline-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental): Low dose or placebo, twice daily
  Interventions: Drug: AZD7325; Drug: Placebo
- 2 (Experimental): Low dose or placebo, once daily
  Interventions: Drug: AZD7325; Drug: Placebo
- 3 (Experimental): Middle dose or placebo, twice daily
  Interventions: Drug: AZD7325; Drug: Placebo
- 4 (Experimental): High dose or placebo, once daily
  Interventions: Drug: AZD7325; Drug: Placebo

INTERVENTIONS:
Drug: AZD7325 — oral capsule, once or twice daily, 7 days
Drug: Placebo — oral capsule, once or twice daily, 7 days

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability after repeated ascending doses of AZD7325 in Japanese healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Japanese subjects

Exclusion Criteria:

* Significant illness, as judged by the investigator, within 2 weeks of Day 1
* Enrollment in another concurrent investigational study or intake of an investigational drug within 4 months prior to the screening visit
* Blood loss in excess of 200 mL within 30 days of Day 1, in excess of 400 mL within 90 days of Day 1, or in excess of 1200 mL within 1 year of Day 1
* Clinically relevant abnormalities in physical examinations, vital signs, clinical chemistry, hematology or urinalysis as judged by the investigator and/or sponsor

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-07; Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of multiple ascending oral doses of AZD7325 compared to placebo in healthy male Japanese subjects by assessment of adverse events, vital signs, physical examinations, laboratory parameters, ECGs and EEG. | Observations/Assessments are made at each visit (Screening visit, Treatment visit (Day 1-Day 9) and Follow-up visit).

SECONDARY OUTCOMES:
To evaluate and characterize the pharmacokinetics of AZD7325 when given orally in multiple ascending doses by assessment of drug concentration in plasma and urine. | Blood and urine samples will be taken before and after study drug administration (up to 48 hours post dose).
To evaluate the effects on VAS, Ataxia assessments and CogState Battery (cognition). | Observations/Assessments are made during the treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Kumagai, MD, PhD, Principal Investigator — Kitasato University East Hospital, Kanagawa, Japan